CLINICAL TRIAL: NCT00141375
Title: An Open-Label Extension to Evaluate the Safety and Efficacy of Pregabalin for Treatment of Chronic Central Neuropathic Pain After Spinal Cord Injury.
Brief Title: To Evaluate Long-Term Safety and Efficacy of Pregabalin in the Treatment of Neuropathic Pain After Spinal Cord Injury.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1008-000-202
Record Dates: First submitted 2005-08-30; First posted 2005-09-01 (Estimated); Last update posted 2008-01-15 (Estimated); Status verified 2008-01

CONDITIONS: Neuropathic Pain
MeSH Terms: conditions — Neuralgia | interventions — Pregabalin

INTERVENTIONS:
Drug: Pregabalin

SUMMARY:
To evaluate long-term safety and efficacy of pregabalin in the treatment of neuropathic pain after spinal cord injury.

ELIGIBILITY:
Inclusion Criteria:

* Must have met the inclusion criteria of the preceding double-blind BID study in central pain following spinal cord injury.
* Must have received study medication under double-blind conditions.

Exclusion Criteria:

* Patients cannot participate if they experienced a serious adverse event during the previous double-blind BID study which was determined to be related to the study medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132
Dates: Start 2002-08; Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Safety and Efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (7):
- Australia (7):
  - Pfizer Investigational Site, Little Bay, New South Wales
  - Pfizer Investigational Site, St Leonards, New South Wales
  - Pfizer Investigational Site, Warrawong, New South Wales
  - Pfizer Investigational Site, Woolloongabba, Queensland
  - Pfizer Investigational Site, Heidelberg, Victoria
  - Pfizer Investigational Site, Shenton Park, Western Australia
  - Pfizer Investigational Site, NSW